CLINICAL TRIAL: NCT06524375
Title: Phase II, Open-label, Prospective Single-arm, Multi-center Clinical Trial to Evaluate if Adding Venetoclax to Patients on Covalent BTKi For 1L CLL Can Achieve Deep Durable Remissions (by UMRD 10^-4) to Allow Off-treatment Period.
Brief Title: A Study to Evaluate the Effect of Venetoclax on Participants Receiving a Covalent Bruton's Tyrosine Kinase Inhibitor (cBTKi) for First-line Chronic Lymphocytic Leukemia (1L CLL) to Achieve Deep Durable Remissions to Allow Off-treatment Period.
Acronym: BRAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML45219
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax Added to cBTKi (Commercially Prescribed) (Experimental): Participants will receive venetoclax, orally, once daily (QD) with a starting ramp-up dose of 20 milligrams (mg) on Day 1 of Cycle 1 (cycle length= 28 days). The dose will increase weekly; thereafter, treatment will continue with venetoclax at the target dose of 400 mg, QD from Day 1 of Cycle 2 up to Day 28 of Cycle 12.
  Participants will continue receiving cBTKi-monotherapy (i.e. ibrutinib or acalabrutinib, or zanubrutinib) as previously prescribed by the investigator according to the prescribing label.
  Interventions: Drug: Venetoclax; Drug: cBTKi Monotherapy

INTERVENTIONS:
Drug: Venetoclax — Venetoclax tablets will be administered as per the schedule specified in the arm.
  Other Names: RO5537382
Drug: cBTKi Monotherapy — Commercially available cBTKi (ibrutinib or acalabrutinib, or zanubrutinib) will be administered in accordance with its prescribing label.

SUMMARY:
The main purpose of the study is to evaluate if adding venetoclax to participants receiving cBTKi for the 1L CLL can achieve deep durable remissions of undetectable measurable residual disease [uMRD < or 10^-4 in peripheral blood (PB)] by end of combination treatment (EOCT) to allow off-treatment period.

The acronym BRAVE stands for Btki Responders to Achieve deep remission (or off-treatment periods) with VEnetoclax.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CLL and currently receiving a stable dose of cBTKi (i.e., ibrutinib, acalabrutinib, or zanubrutinib) for at least 6 months for 1L treatment with a response of at least a PR per iwCLL criteria
2. Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to (</=) 2
3. Adequate renal and liver function

Exclusion Criteria:

1. Prior B-cell lymphoma (Bcl-2) inhibitor therapy
2. Anti-cluster of differentiation 20 (CD20) therapy within the month prior to screening
3. Progressive or stable disease on cBTKi
4. Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (Richter's transformation or pro-lymphocytic leukemia)
5. History of cardiomyopathy
6. Hypersensitivity to venetoclax or to any of the excipients (e.g., trehalose)
7. Clinically significant cardiovascular disease
8. Active bleeding or history of bleeding diathesis
9. Pregnant women and nursing mothers
10. Uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-02-08 (Estimated); Study Completion 2028-02-08 (Estimated)

PRIMARY OUTCOMES:
Undetected Minimal Residual Disease at 10^-4 (uMRD4) PB Rates at EOCT | Cycle 12 Day 28 (Cycle length= 28 Days)
  uMRD4 will be assessed using next generation sequencing (NGS) (sensitivity 10^-4) from PB.

SECONDARY OUTCOMES:
CR/CRi Rate at EOCT as Determined by the Investigator According to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines | Up to approximately 12 months
  Complete response (CR) / complete response with incomplete recovery of the bone marrow (CRi) rate is defined as the percentage of participants with a CR or CRi, as determined by the investigator according to the iwCLL.
Partial Response (PR) Rate at EOCT as Determined by the Investigator According to iwCLL Guidelines | Up to approximately 12 months
  PR rate is defined as the percentage of participants with a PR, as determined by the investigator according to the iwCLL.
Overall Response Rate (ORR) at EOCT as Determined by the Investigator According to iwCLL Guidelines | Up to approximately 12 months
  ORR is defined as the percentage of participants with a CR/CRi or PR, as determined by the investigator according to the iwCLL.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 24 months
  Adverse events including adverse events of special interest (AESIs) and SAEs will be collected as part of this study at baseline and every clinical visit, until 30 days after the final dose of study treatment.
Number of Participants Who Withdrew Prematurely from the Study | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (21):
  - Highlands Oncology Group, Springdale, Arkansas
  - Rocky Mountain Cancer Centers (Aurora) - USOR, Aurora, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - Mission Blood and Cancer - MercyOne Cancer Center, Des Moines, Iowa
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Dana-Farber Cancer Institute - Hematologic Oncology Treatment Center, Boston, Massachusetts
  - Nebraska Cancer Specialists St Francis - Grand Island, Grand Island, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - San Juan Oncology Associates, PC, Farmington, New Mexico
  - Oncology Hematology Care Inc - Cincinnati - USOR, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Tennessee Oncology, PLLC - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology - Midtown, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing